CLINICAL TRIAL: NCT00949130
Title: A Multicenter,Investigator-blinded,Randomized, Comparative Study to Evaluate the Efficacy and Safety of Oral NXL103 Versus Oral Linezolid in the Treatment of Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Brief Title: Comparative Study of NXL103 Versus Linezolid in Adults With Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novexel Inc (Industry)
Responsible Party: Dr. Michael Kuligowski, Director of Clinical Research, Novexel Inc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NXL103/2002
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Acute Bacterial Skin and Skin Structure Infections
MeSH Terms: interventions — flopristin, linopristin drug combination; Linezolid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NXL103 (Experimental): BID for 7-14 days orally
  Interventions: Drug: NXL103
- Linezolid (Active Comparator): BID for 7-14 days orally
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: NXL103 — BID for 7-14 days
  Arms: NXL103
Drug: Linezolid — BID for 7-14 days
  Arms: Linezolid

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of oral NXL103 vs. established treatment of acute bacterial infection in adults.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute bacterial skin and skin structure infection (ABSSSI) with at least 3 signs or symptoms

Exclusion Criteria:

* Uncomplicated acute bacterial skin and skin structure infections
* ABSSSI suspected or proven to be due to Gram negative and/or anaerobic pathogens
* Pregnant or lactating women
* Inadequately controlled diabetes mellitus
* Inadequately controlled arterial hypertension
* Moderate-to-severe renal impairment
* Moderate-to-severe liver disease
* Conditions associated with immunodeficiency
* Known hypersensitivity or any contraindication for the use of any of the 2 study drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Clinical response at the early follow-up visit (Test of cure) | 7 days post therapy

SECONDARY OUTCOMES:
Clinical outcome at the late follow-up visit | 21 days post therapy
Clinical outcome at the end of treatment | 10-14 days therapy
Microbiological outcome at the early follow-up visit (Test of cure) | 7 days post-therapy
Safety Profiles (safety and tolerability) | throughout the study
Population pharmacokinetic profile of the experimental study drug | Day 1-5 while on study drug

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuligowski, MD, Study Director — Novexel Inc
Locations (15):
- United States (11):
  - Sharp Chula Vista Research Office, Chula Vista, California
  - Fountain Valley Regional Hospital and Medical Center, Fountain Valley, California
  - Sharp Grossmont Research Office, La Mesa, California
  - Tri-City Oceanside Office, Oceanside, California
  - Southeast Regional Research Group, Columbus, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - Idaho Falls Infectious Diseases, Idaho Falls, Idaho
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Infectious Diseaes MPLS-LTD, Minneapolis, Minnesota
  - Mercury Street Medical Group, Butte, Montana
  - RPS Infectious Diseases, West Reading, Pennsylvania
- Guatemala (4):
  - Roosevelt Hospital, Guatemala City
  - UNICAR, Guatemala City
  - Military Health Center, Guatemala City
  - Private Hospital, Quetzaltenango